CLINICAL TRIAL: NCT05730556
Title: Remote Electrical Neuromodulation for Acute Procedural Pain in Chronic Migraine Patients Receiving onabotulinumtoxinA
Brief Title: A Study of Remote Electrical Neuromodulation for Acute Procedural Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enough data was collected to demonstrate device efficacy at interim analysis
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amaal J. Starling, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 22-011180
Record Dates: First submitted 2023-02-06; First posted 2023-02-16 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-09

CONDITIONS: Chronic Migraine
Keywords: OnabotulinumtoxinA (Botox) injections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Electrical Neuromodulation, Then Sham (Experimental): Subjects will first have the Nerivio ® applied 20 minutes prior to clinical care onabotulinumtoxinA (Botox) injection, and continue to wear the device for a total of 40 to 45 minutes at week 12. Subjects will then have the sham device applied 20 minutes prior to clinical care onabotulinumtoxinA (Botox) injection, and continue to wear the device for a total of 40 to 45 minutes at week 24.
  Interventions: Device: Nerivio ®; Device: Sham
- Sham, Then Electrical Neuromodulation (Experimental): Subjects will first have the sham device applied 20 minutes prior to clinical care onabotulinumtoxinA (Botox) injection, and continue to wear the device for a total of 40 to 45 minutes at week 12. Subjects will then have the Nerivio ® applied 20 minutes prior to clinical care onabotulinumtoxinA (Botox) injection, and continue to wear the device for a total of 40 to 45 minutes at week 24.
  Interventions: Device: Nerivio ®; Device: Sham

INTERVENTIONS:
Device: Nerivio ® — Non-invasive wearable, remote electrical neuromodulation (REN) device controlled by a smartphone application worn on an armband on the upper arm.
Device: Sham — Electrical stimulation to mimic study treatment intervention

SUMMARY:
The purpose of this study is to assess the effectiveness of using remote electrical neuromodulation, using the Nerivio ® device, to relieve pain associated with receiving onabotulinumtoxinA (Botox) injections for chronic migraine prevention.

ELIGIBILITY:
Inclusion Criteria:

* Meet the criteria for 1.3 chronic migraine based on ICHD3 criteria.
* Currently receiving onabotulinumtoxinA per PREEMPT protocol for the treatment of chronic migraine.
* Patient is willing and able to comply with the protocol to the satisfaction of the investigator.
* Patient has the capacity to provide written, informed consent for themselves.

Exclusion Criteria:

* Participants with an active implanted electrical and/or neurostimulator device (e.g., cardiac pacemaker, cochlear implant).
* Participants with congestive heart failure (CHF), severe cardiac or cerebrovascular disease.
* Participants with uncontrolled epilepsy.
* Pregnant, trying to get pregnant or breastfeeding female participants.
* Subjects participating in any other interventional clinical study.
* Participants with other significant pain, medical or psychological problems that in the opinion of the investigator may confound the study assessments.
* Participants who have previous experience with the device.
* Patients with cranial deformities, prior cranial surgeries with violation of the calvarium, or shunt placement.
* Patients receiving concurrent nerve blocks or trigger point injections within the same visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amaal Starling, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 80 participants were consented to the study and of those 80 participants, 20 were withdrawn prior to randomization.
Groups:
- Electrical Neuromodulation, Then Sham: Subjects first had the Nerivio ® applied 20 minutes prior to clinical care onabotulinumtoxinA (Botox) injection, and continued to wear the device for a total of 40 to 45 minutes at week 12. Subjects then had the sham device applied 20 minutes prior to clinical care onabotulinumtoxinA (Botox) injection, and continued to wear the device for a total of 40 to 45 minutes at week 24.
  Nerivio ®: Non-invasive wearable, remote electrical neuromodulation (REN) device controlled by a smartphone application worn on an armband on the upper arm.
  Sham: Electrical stimulation to mimic study treatment intervention
- Sham, Then Electrical Neuromodulation: Subjects first had the sham device applied 20 minutes prior to clinical care onabotulinumtoxinA (Botox) injection, and continued to wear the device for a total of 40 to 45 minutes at week 12. Subjects then had the Nerivio ® applied 20 minutes prior to clinical care onabotulinumtoxinA (Botox) injection, and continued to wear the device for a total of 40 to 45 minutes at week 24.
  Nerivio ®: Non-invasive wearable, remote electrical neuromodulation (REN) device controlled by a smartphone application worn on an armband on the upper arm.
  Sham: Electrical stimulation to mimic study treatment intervention
Period: First Intervention
Arm/Group | Electrical Neuromodulation, Then Sham | Sham, Then Electrical Neuromodulation
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Electrical Neuromodulation, Then Sham | Sham, Then Electrical Neuromodulation
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Electrical Neuromodulation, Then Sham | Sham, Then Electrical Neuromodulation | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (12.2) | 44.5 (15.0) | 48.0 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 23 | 49
  Male | 4 | 7 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity Measured by Visual Analog Scale (VAS)
Description: Measured by VAS values reported by participants using the 100-mm Visual Analogue Scale (VAS). The VAS line will be 100 mm long with no intermediate delineations. Each end will be marked with "no pain" on the left, and "worst possible pain" on the right. Participants will identify their pain level by indicating a point on the line between each end. That point will be measured from the "No pain" end, and the number of millimeters will be reported as the pain score. Scores can range from 0 to 100, with higher score indicating worse pain.
Time Frame: Baseline, Week 12, Week 24
Population: Seven (7) participants in the Electrical Neuromodulation, Then Sham arm and Eight (8) participants in Sham, Then Electrical Neuromodulation arm did not have Week 24 data as the trial was stopped early as the stopping rule for efficiency was reached in the interim analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electrical Neuromodulation, Then Sham | Sham, Then Electrical Neuromodulation
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline Pre-Procedure | 23.0 (26.3) | 32.9 (24.8)
  Baseline Intra-Procedure | 52.5 (19.6) | 58.3 (24.2)
  Baseline Post-Procedure | 59.9 (22.1) | 62.0 (25.2)
  Week 12 Pre-Procedure | 21.2 (23.3) | 27.0 (23.7)
  Week 12 Intra-Procedure | 37.2 (19.3) | 60.7 (20.6)
  Week 12 Post-Procedure | 38.7 (19.7) | 64.7 (21.5)
  Week 24 Pre-Procedure: number analyzed (Participants) | 23 | 22
  Week 24 Pre-Procedure | 19.2 (24.7) | 25.7 (20.3)
  Week 24 Intra-Procedure: number analyzed (Participants) | 23 | 22
  Week 24 Intra-Procedure | 50.4 (20.5) | 44.5 (22.8)
  Week 24 Post-Procedure: number analyzed (Participants) | 23 | 22
  Week 24 Post-Procedure | 54.6 (23.4) | 46.6 (25.3)

2. Secondary Outcome: Presence of Post-procedural Headache
Description: Number of subjects to report the presence of post-procedural headache, defined as a headache that lasts for 4 hours or more and is at least moderate in severity or during which abortive medications are used to treat the patient's head pain.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Electrical Neuromodulation, Then Sham | Sham, Then Electrical Neuromodulation
Number analyzed (Participants) | 30 | 30
Participants
  Baseline | 12 | 11
  Week 12 | 4 | 20
  Week 24: number analyzed (Participants) | 23 | 22
  Week 24 | 9 | 4

3. Secondary Outcome: Adverse Events
Description: Number of adverse events reported
Time Frame: 24 weeks
Measure: Number; unit: events
Groups:
- Electrical Neuromodulation: Subjects had the Nerivio ® applied 20 minutes prior to clinical care onabotulinumtoxinA (Botox) injection, and continued to wear the device for a total of 40 to 45 minutes.
  Nerivio ®: Non-invasive wearable, remote electrical neuromodulation (REN) device controlled by a smartphone application worn on an armband on the upper arm.
- Sham, Then Electrical Neuromodulation: Subjects had the sham device applied 20 minutes prior to clinical care onabotulinumtoxinA (Botox) injection, and continued to wear the device for a total of 40 to 45 minutes.
  Sham: Electrical stimulation to mimic study treatment intervention
Arm/Group | Electrical Neuromodulation | Sham, Then Electrical Neuromodulation
Number analyzed (Participants) | 60 | 60
events | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of informed consent through study completion, approximately 24 weeks
Groups:
- Sham: Subjects had the sham device applied 20 minutes prior to clinical care onabotulinumtoxinA (Botox) injection, and continued to wear the device for a total of 40 to 45 minutes.
  Sham: Electrical stimulation to mimic study treatment intervention
Arm/Group | Electrical Neuromodulation | Sham
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

LIMITATIONS AND CAVEATS:
This study was terminated early as enough data was collected at interim analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/56/NCT05730556/Prot_SAP_000.pdf